CLINICAL TRIAL: NCT05221086
Title: Urdu Version of The ProFitMap-neck - Reliability and Validity of a Questionnaire for Measuring Symptoms and Functional Limitations in Chronic Neck Pain
Brief Title: Urdu Version Of ProFitMap-Neck Questionnaire In Population With Chronic Neck Pain A Reliability And Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00260
Record Dates: First submitted 2022-02-01; First posted 2022-02-02 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Chronic Neck Pain
Keywords: Urdu Version of ProFitMap-neck; Non-specific Chronic Neck Pain; Psychometric Properties; Validity; Functional Limitations; Reliability

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to translate or culturally adapt ProFitMap-neck into Urdu language and to investigate the reliability and validity of the ProFitMap-neck in Pakistani population having chronic neck pain. Also check it's correlation with Neck Disability Index.

DETAILED DESCRIPTION:
As with prior suggestions, the English version of the ProFitMap-neck will be translated and culturally modified.In population having Chronic Neck Pain ProFitMap-neck will be distributed among one hundred and thirty six participants selected by a convenience sampling technique based on pre-defined inclusion and exclusion criteria.The questionnaire will be filled out by two observers on the same day to examine inter and intra-observer reliability of the final ProFitMap-neck and neck disability index. For the inter-observer evaluation, there will be a 2 hour delay between the first and second application. After 7 days, observer-1 will conduct a third assessment (re-testing) for intra-observer evaluation.The Statistical Package of Social Sciences program will be used to examine the data.

ELIGIBILITY:
Inclusion Criteria

Non-specific chronic neck pain Age 18-65 years Neck pain that isn't caused by a traumatic event

Exclusion Criteria

Neck pain due to any type of surgery Neck pain as a result of an injury Neck pain due to broken bone or dislocation Rheumatological issues Pregnant women Any Cardiovascular disorders Any Neurological problems Cord compression Insufficiency of the vertebrobasilar artery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pakistani Population with non-specific Chronic Neck Pain.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
ProFitMap-Neck Questionnaire | 1st day
  The functional limitation scale (function index) and the symptom scale (often and much) are the two original ProFitMap-neck measures,each with 20 and 27 items, respectively. There are six response options for each item, which fall into the following categories. The function index ranges from ''very good, no problems, very satisfying, very likely" to ''very awful, extremely difficult/impossible, extremely dissatisfying, extremely unlikely", Symptom scale with intensity index (how much) ranging from ''nothing/nothing at all" to ''nearly unbearable/ terrible, all/maximally"; The frequency index (how often) ranges from ''never/very seldom" to ''very often/always" on the symptom scale.The index values are scaled from 0 to 100. Higher ratings indicate improved function/health. The intensity index and the frequency index are two different types of indexes.
Neck Pain Disability Index | 1st day
  The Neck Pain Disability Index assesses the severity of neck pain symptoms and its impact on daily life. It has ten sections that cover pain intensity, attention/focus, headaches, and daily activities. The items include six response options ranging from no disability (0) to total disability (5), giving a total score of 0 to 50.The Neck Disability index was normalized from 0 to 100 in this study, with higher scores indicating more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No